CLINICAL TRIAL: NCT05084638
Title: AGNOS: An 18-month, Open-label, Multi-Center Study to Assess the Effect of Ofatumumab 20mg SC Monthly in Treatment Naïve, Very Early Relapsing Remitting Multiple Sclerosis Patients Benchmarked Against Healthy Controls on Select Outcomes.
Brief Title: Study to Assess the Effect of Ofatumumab in Treatment Naïve, Very Early RRMS Patients Benchmarked Against Healthy Controls.
Acronym: AGNOS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COMB157GUS10
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Relapse Remitting Multiple Sclerosis
Keywords: early relapsing multiple sclerosis; ofatumumab; healthy control; treatment naïve; young adult population; MS-related disability; biomarker; MRI
MeSH Terms: interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ofatumumab (Experimental): Ofatumumab will be provided in an autoinjector for subcutaneous administration. Dosing regimen for this study is an initial dose of 20mg at Baseline/Week 0, followed by Week 1, 2 and every month thereafter, beginning at Week 4 (Month 1) until Month 18. There will be an optional extension of dosing through month 30.
  Interventions: Drug: Ofatumumab
- Healthy Control (No Intervention): Healthy Control arm will be age- and sex-matched subjects (to the ofatumumab treated arm) and will not receive a study treatment.

INTERVENTIONS:
Drug: Ofatumumab — 20mg subcutaneous injection
  Other Names: OMB157
  Arms: Ofatumumab

SUMMARY:
This study will evaluate the impact of ofatumumab in Relapsing Remitting Multiple Sclerosis (RRMS) participants that are very early in the course of their disease using clinical and magnetic resonance imaging (MRI) outcomes. The study will also assess changes in disease using monitoring techniques including digital biometric device use, biomarker analysis and non-conventional MRI. Select outcomes in the ofatumumab treated group will be compared to a group of Healthy participants to determine if there are similarities between the groups after the patients with MS undergo treatment with ofatumumab.

DETAILED DESCRIPTION:
The study is an open-label, multi-center, prospective 18-month study in 118 MS participants with early RRMS (defined as within 6 months of diagnosis of clinically definite RRMS) and who are treatment naïve. It is designed to determine if RRMS participants treated with 20 mg subcutaneous monthly ofatumumab during the earliest part of their disease will benefit from the use of ofatumumab as their first disease modifying therapy. Additionally, RRMS patients will be compared to age- and sex-matched healthy participants (n=50) for select outcomes to observe similarities and differences between the groups.

After giving consent, participants will have a 28-day screening/qualification period. If they qualify to continue, they will start study measures including assessments of clinical and magnetic resonance imaging (MRI) metrics and use of a digital monitoring watch. Additionally, samples will be collected for laboratory and biomarker analysis. RRMS participants will begin treatment with ofatumumab for the next 18 months. Healthy participants will undergo similar assessments; however they will not receive any treatment during the course of the study. Over the 18 months, participants will have regular clinical visits with assessments and sample collection. After 18 months in the trial, participants in both groups will have the option to enter into a 12-month extension (up to 30 months total in study) to collect further information on long-term clinical and MRI outcomes.

ELIGIBILITY:
Key Inclusion Criteria:

Participants eligible for inclusion in this study must meet all of the following criteria:

1. Signed informed consent must be obtained prior to participation in the study
2. Age 18-35 years

   Patients in the healthy control arm eligible for inclusion must fulfill the following criteria:
3. Able to obtain MRI (HC with abnormal MRI at Screening will be excluded) and use wearable device
4. Able to provide blood sample (no CSF will be collected in HC)

   Patients in the ofatumumab-treated arm eligible for inclusion must fulfill the following criteria:
5. Diagnosis of RRMS per McDonald Criteria (2010/2017)
6. Within 6 months of diagnosis of clinically definite MS (CDMS)
7. EDSS 0-3.0 (Inclusive)
8. Treatment-naïve to MS DMT
9. Able to obtain MRI and attend study visits at sites
10. Able to use wearable device
11. Able to provide blood sample (and CSF for sub-group n=15)

Key Exclusion Criteria:

Participants in the healthy control arm meeting any of the following criteria are not eligible for inclusion in this study:

1. Confounding medical condition as determined by the investigator

   RRMS patients fulfilling any of the following exclusion criteria are not eligible for inclusion in this study:
2. Diseases other than multiple sclerosis responsible for the clinical or MRI presentation
3. Patients with neuromyelitis optica, Radiologic/ Clinically Isolated Syndrome, Secondary Progressive or Primary Progressive MS diagnosis
4. Use of experimental or investigational drugs for MS
5. Previous use of Disease Modifying Therapy (DMT) or chemotherapeutic medications for MS
6. Relapse between screening and Baseline visits
7. Known sensitivity to gadolinium; patients with chronic, severe kidney disease
8. Known history of hypersensitivity to any of the study treatments or its excipients or to drugs of similar chemical classes
9. CNS anomalies that are better accounted for by another disease process or MRI anomalies causing clinically apparent impairments
10. Known active malignancies
11. Pregnant or nursing (lactating) women
12. Females of childbearing potential (all women physiologically capable of becoming pregnant) should use effective contraception while receiving ofatumumab and for 6 months after the last treatment of ofatumumab
13. Patients with an active chronic disease (or stable but treated with immune therapy) of the immune system other than MS or with immunodeficiency syndrome
14. Patients with active infections including systemic bacterial, viral (including SARS-CoV-2/COVID-19) or fungal infections, or known to have AIDS or to test positive for HIV antibody at Screening
15. Patients with neurological findings consistent with Progressive Multifocal Leukoencephalopathy (PML), or confirmed PML
16. Patients with IgG or IgM levels below LLN at Screening
17. Patients that have received any live or live-attenuated vaccines within 4 weeks prior to first dose of study drug administration
18. Patients at risk of developing or having reactivation of hepatitis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2026-02-16 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving NEDA-3 (No Evidence of Disease Activity-3) | Month 6 to month 18
  A participant is considered as achieved NEDA-3 if the participant has not had a clinical relapse (recurrence of a disease activity after a recovery), has not had an increase in disability and has no new radiological MRI activity (no new occurrences of contrast-enhancing lesions) during study Months 6 to 18.

SECONDARY OUTCOMES:
Number of relapses | Baseline to Month 18 and 30
  Relapses are recurrences of a disease activity after a recovery. A confirmed MS relapse is one accompanied by a clinically relevant change in the EDSS performed by the EDSS Rater, i.e. an increase of at least 0.5 points on the EDSS score, or an increase of 1 point on two functional scores (FSs) or 2 points on one FS, excluding changes involving bowel/bladder or cerebral FS compared to the previous available rating (the last EDSS rating that did not occur during a relapse). Confirmation of MS relapse based on these definitions will be done centrally.
Number of participants that were 3-month Disability Worsening-free | Baseline up to Month 18 and 30
  No increase or worsening of disability over a period of 3 months or more
Number of participants with NEDA (No Evidence of Disease Activity) - Clinical | Month 6 to Month 18
  A participant is considered as achieved NEDA-Clinical if the participant has not had a clinical relapse (recurrence of a disease activity after a recovery).
Number of participants with NEDA (No Evidence of Disease Activity) - Radiological | Month 6 to Month 18
  A participant is considered as achieved NEDA-radiological if the participant has has no new radiological MRI activity (no new occurrences of contrast-enhancing lesions) during study Months 6 to 18.
Change from Baseline in Gd+ lesion count | Baseline to Month 18 and 30
  Change in the number of gadolinium enhancing lesions will be measured by Magnetic Resonance Imaging (MRI). Each MRI scan will be previewed by a local neuroradiologist. The quality of each scan performed will be assessed by a central MRI reading center.
Change from Baseline in Gd+ lesion volume | Baseline to Month 18 and 30
  Change in size of gadolinium enhancing lesions will be measured by Magnetic Resonance Imaging (MRI). Each MRI scan will be previewed by a local neuroradiologist. The quality of each scan performed will be assessed by a central MRI reading center.
Change from Baseline in new/enlarging T2 lesion count | Baseline to Month 18 and 30
  Change in the number of new/enlarging T2 lesions will be measured by Magnetic Resonance Imaging (MRI). Each MRI scan will be previewed by a local neuroradiologist. The quality of each scan performed will be assessed by a central MRI reading center.
Change from Baseline in T2 lesion volume | Baseline to Month 18 and 30
  Change in size of T2 lesions will be measured by Magnetic Resonance Imaging (MRI). Each MRI scan will be previewed by a local neuroradiologist. The quality of each scan performed will be assessed by a central MRI reading center.
Change from Baseline for NeuroQOL | Baseline to Month 18 and 30
  The NeuroQOL is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The following domains will be measured.
  Physical Health, Mental Health, Social Health. Scales can be scored by summing the values of the response to each item to develop a total raw score.
Change from Baseline for Patient Determined Disease Steps (PDDS) | Baseline to Month 18 and 30
  The PDDS is a standardized rating scale which is a self-assessment scale of functional disability in multiple sclerosis patients primarily based on ambulation. The questionnaire contains 1 question which is scored ranging from 0 (normal) to 8 (bedridden). A score of 0 to 2 indicates mild disability; a score of 3 to 5 indicates moderate disability; a score of 6 to 8 indicates severe disability.
Brain volume loss (BVL) assessment (whole brain and regional) | Month 6 to Month 18 and 30
  Brain volume loss is a marker of progressive loss of brain structure and function. It is a predictor of disability progression. Evaluate the effect of ofatumumab vs healthy controls on 1) whole brain and regional atrophy measured at month 18/30 after re-baseline at 6 months; and 2) regional atrophy measured 18/30 months from Baseline
Number of participants with treatment emergent adverse events | Baseline up to approximately Month 30
  Adverse event monitoring should be continued following the last dose of study treatment until B cells are repleted. Repletion is defined as a concentration > the participant's baseline value or > the lower limit of normal, whichever is observed first. Other safety assessments (physical exam, vital signs, etc) that meet the definition of an adverse event or are considered clinically relevant by the investigator will be reported as an adverse event.
Change from Baseline in new unenhancing T1 lesion number | Baseline to Month 18 and 30
  Change in the number of new unenhancing T1 lesions will be measured by Magnetic Resonance Imaging (MRI). Each MRI scan will be previewed by a local neuroradiologist. The quality of each scan performed will be assessed by a central MRI reading center.
Change from Baseline in T1 unenhancing lesion volume | Baseline to Month 18 and 30
  Change in the size of T1 unenhancing lesions will be measured by Magnetic Resonance Imaging (MRI). Each MRI scan will be previewed by a local neuroradiologist. The quality of each scan performed will be assessed by a central MRI reading center.

CONTACTS AND LOCATIONS:
Locations (36):
- United States (35):
  - MD First Research, Chandler, Arizona
  - Barrow Neurological Clinics at St Josephs Hospital and MC, Phoenix, Arizona
  - Arizona Neuroscience Research LLC, Phoenix, Arizona
  - Keck School of Medicine, Los Angeles, California
  - Lundquist Inst BioMed at Harbor, Torrance, California
  - Regina Berkovich MD PhD Inc, West Hollywood, California
  - UC Health Neuroscience Ctr, Aurora, Colorado
  - MedStar Health, Washington D.C., District of Columbia
  - Neurology of Central FL Res Ctr, Altamonte Springs, Florida
  - First Choice Neurology, Boca Raton, Florida
  - Univ of Florida College of Medicine, Gainesville, Florida
  - Neurology Associates PA, Maitland, Florida
  - Orlando Health Clinical Trials, Orlando, Florida
  - Emerald Coast Neurology, Pensacola, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - University Of South Florida, Tampa, Florida
  - Shepherd Center, Atlanta, Georgia
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Renown Institute for Neurosciences, Reno, Nevada
  - Neuroscience Institute at Hackensack, Hackensack, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Velocity Clinical Research, Raleigh, North Carolina
  - Neurology Diagnostics Inc, Dayton, Ohio
  - Multiple Sclerosis Center of Excellence of OMRF, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Sibyl Wray MD Neurology PC, Knoxville, Tennessee
  - Univ of Texas Southwest Med Center, Dallas, Texas
  - UT Health Science Center, Houston, Texas
  - Lonestar Neurology of San Antonio, San Antonio, Texas
  - Evergreen Health Multiple Sclerosis Center, Kirkland, Washington
  - MultiCare Neuroscience Center of Washington, Tacoma, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Caribbean Center for Clinical Research, Inc, Guaynabo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com